CLINICAL TRIAL: NCT00531687
Title: Phase II Trial of Paclitaxel, Gemcitabine and Cisplatin in Patients With Relapsing Germ Cell Cancer
Brief Title: Trial of Paclitaxel, Gemcitabine and Cisplatin in Patients With Relapsing Germ Cell Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gedske Daugaard, Associate professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Relapse testis cancer 2007
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Testicular Cancer
Keywords: relapse
MeSH Terms: conditions — Testicular Neoplasms; Recurrence | interventions — Paclitaxel; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GCT (Other): cisplatin Paclitaxel gemcitabine
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 175 mg/m2 day 1 (3 hour infusion)
  Repeat at 21-day intervals for 4 cycles if toxicity is acceptable. If necessary more than 4 cycles can be administered.
  Other Names: taxol
Drug: Cisplatin — cisplatin 50 mg/m2 day 1 and 2
  Repeat at 21-day intervals for 4 cycles if toxicity is acceptable. If necessary more than 4 cycles can be administered.
Drug: Gemcitabine — gemcitabine 1000mg/m2 days 1 and 8 (in a 30 minute infusion)
  Repeat at 21-day intervals for 4 cycles if toxicity is acceptable. If necessary more than 4 cycles can be administered
  Other Names: Gemzar

SUMMARY:
Study Objectives:

Primary objective

* The primary objective of this study is to investigate the combination of cisplatin/gemcitabine/paclitaxel, with respect to complete remission in patients with germ cell tumours previously treated with BEP.

Secondary Objectives

* Overall survival
* Progression free survival
* Response rates (RECIST)
* Duration of response
* To investigate the safety of paclitaxel, gemcitabine and cisplatin in patients previously treated with BEP

DETAILED DESCRIPTION:
not relevant

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed germ cell tumor (seminoma or non-seminoma) with measurable metastatic disease either by radiography (at a site which has previously not been irradiated) or elevation of alpha fetoprotein (AFP) and/or elevation of beta-human chorionic gonadotropin (beta-HCG);
* Patient previously treated with standard BEP (3 or 4 cycles) with relapse 1 months or more after favorable response on previous chemotherapy (CR or PR)
* Male
* Age greater than or equal to 18 years;
* Performance status 0,1,2 or 3
* WBC > 3000 mill/l, ANC > 1500 mill/l, platelet count > 100.000 mill/l; serum bilirubin < 1.5 x the upper limit of normal;
* Adequate renal function (Glomerular Filtration Rate (GFR) >60 ml/min). GFR will be assessed by direct measurement (EDTA clearance or creatinine clearance)
* signed informed consent;

Exclusion Criteria:

* Uncontrolled active severe clinical infection (CTC grade 3 or 4).
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator), including expected difficulty of follow-up related to mental disorders.
* Grade 2 or greater peripheral neuropathy according to the CTC, version 3.0.
* Second malignancy other than basal or squamous cell skin cancer.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-09; Primary Completion 2012-02 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Primary objective · The primary objective of this study is to investigate the combination of cisplatin/gemcitabine/paclitaxel, with respect to complete remission in patients with germ cell tumours previously treated with BEP. · · | December 2010

SECONDARY OUTCOMES:
Secondary Objectives · Overall survival | 5 years
Secondary Objectives · Progression free survival | 5 years
Secondary Objectives · Response rates (RECIST) | 5 years
Secondary Objectives · Duration of response | 5 years
Secondary Objectives · To investigate the safety of paclitaxel, gemcitabine and cisplatin in patients previously treated with BEP | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gedske Daugaard, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Oncology 5073, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No